CLINICAL TRIAL: NCT04384770
Title: Magnetic Resonance Imaging-Guided Stereotactic Body Radiotherapy for Prostate Cancer (Mirage): A Phase III Randomized Trial
Brief Title: CT-guided Stereotactic Body Radiation Therapy and MRI-guided Stereotactic Body Radiation Therapy for Prostate Cancer, MIRAGE Study
Status: Active, not recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-000328; NCI-2020-02911 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (CT-SBRT): Patients undergo 5 fractions of CT-guided SBRT over 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: CT-guided Stereotactic Body Radiation Therapy; Other: Questionnaire Administration
- Group II (MRI-SBRT): Patients undergo 5 fractions of MRI-guided SBRT over 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: MRI-guided Stereotactic Body Radiation Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: CT-guided Stereotactic Body Radiation Therapy — Undergo CT-guided SBRT
  Other Names: Computed Tomography-Guided Stereotactic Body Radiation Therapy; CT-guided SBRT
  Groups: Group I (CT-SBRT)
Radiation: MRI-guided Stereotactic Body Radiation Therapy — Undergo MRI-guided SBRT
  Other Names: Magnetic Resonance Imaging-guided Stereotactic Body Radiation Therapy; MR-guided SBRT; MRI-guided SBRT
  Groups: Group II (MRI-SBRT)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies compares CT-guided stereotactic body radiation therapy and MRI-guided stereotactic body radiation therapy (SBRT) in treating prostate cancer. Image-guided SBRT is a standard treatment for prostate cancer, which combines imaging of the cancer within the body with the delivery of therapeutic radiation doses produced on a linear accelerator machine. Imaging modalities for image-guided SBRT can be either computed tomography imaging (CT), magnetic resonance imaging (MRI), or a combination of the two. This research is being done to help determine whether there are benefits to MRI-guidance over CT-guidance in patients who are receiving the same radiation dose by SBRT to treat prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether (MRI)-guided stereotactic body radiotherapy (SBRT) improves acute physician-scored genitourinary (GU) toxicity when compared with standard computed tomography (CT)-guided SBRT for prostate cancer (PCa).

SECONDARY OBJECTIVES:

I. To determine whether there are differences in acute grade >= 2 gastrointestinal (GI) toxicity as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale, following MRI-guided SBRT versus CT-guided SBRT.

II. To determine whether there are differences in 5-year cumulative incidences of late grade >= 2 GU and GI physician-reported toxicity, following MRI-guided SBRT versus CT-guided SBRT.

III. To quantify the temporal changes in patient-reported quality of life (QOL) outcomes, as assessed by the Expanded Prostate Cancer Index-26 (EPIC-26), International Prostate Symptom Scores (IPSS), and Sexual Health Inventory for Men (SHIM) QOL indices, following MRI-guided SBRT.

IV. To determine whether there are differences in 5-year biochemical recurrence-free survival (BCRFS) following MRI-guided SBRT.

V. To observe the proportion of SBRT fractions for which on-line adaptive radiotherapy is required due to changes in organ-at-risk anatomy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo 5 fractions of CT-guided SBRT over 14 days in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients undergo 5 fractions of MRI-guided SBRT over 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, clinical localized adenocarcinoma of the prostate
* No evidence of disease beyond the prostate and/or seminal vesicles (i.e., no suspicious pelvic lymph nodes or presence of metastatic disease outside the pelvis)
* Staging workup as recommended by the National Comprehensive Cancer Network (NCCN) on the basis of risk grouping:

  * Low risk: No staging workup required
  * Favorable intermediate-risk: CT abdomen/pelvis if Memorial Sloan Kettering Cancer Center (MSKCC) nomogram predicts >10% probability of lymph node involvement
  * Unfavorable intermediate-risk: technetium bone scan, CT abdomen/pelvis if MSKCC nomogram predicts >10% probability of lymph node involvement
  * High-risk: technetium bone scan, CT abdomen/pelvis if MSKCC nomogram predicts >10% probability of lymph node involvement
  * Advanced imaging studies (i.e. prostate-specific membrane antigen positron emission tomography [PSMA PET] and axumin scan) can supplant a bone scan if performed first
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with any evidence of distant metastases. Note, evidence of lymphadenopathy below the level of the renal arteries can be deemed loco regional per the discretion of the investigator
* Prior cryosurgery, high intensity focused ultrasound (HIFU) or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia
* Contraindications to MRI, including:

  * Electronic devices such as pacemakers, defibrillators, deep brain stimulators, cochlear implants;
  * Metallic foreign body in the eye or aneurysm clips in the brain;
  * Severe claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving stereotactic body radiation therapy for the treatment of prostate cancer at the University of California, Los Angeles
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute grade >= 2 genitourinary (GU) physician-reported toxicity | 90 days after stereotactic body radiation therapy (SBRT)
  Will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale.

SECONDARY OUTCOMES:
Incidence of acute grade >= 2 gastrointestinal (GI) toxicity | 90 days after SBRT
  Will be assessed by the CTCAE version 4.03 scale and rates will be reported descriptively
Incidences of late grade >= 2 GU toxicity | Up to 5 years
  Will be assessed by the CTCAE version 4.03 scale and analyzed using a cumulative incidence framework.
incidences of late grade >= 2 GI toxicity | Up to 5 years
  Will be assessed by the CTCAE version 4.03 scale and analyzed using a cumulative incidence framework.
Patient-reported quality of life (QOL) outcomes | Up 5 years
  For the Expanded Prostate Cancer Index- 26 (EPIC-26) instrument, these will be represented by changes from baseline in the urinary incontinence, urinary obstruction, bowel, sexual function, and hormone/vitality domains. Changes will be analyzed with respect to whether they represent minimally important differences. For the International Prostate Symptom Score (IPSS) and Sexual Health Inventory for Men (SHIM) instruments, the numerical change from baseline, as well as the raw score at any given timepoint, will be extracted.
Biochemical recurrence-free survival (BCRFS) | 5 years
  Will be estimated using the Kaplan-Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum)., with biochemical recurrence (BCR) defined as serum PSA levels that are 2 ng/mL higher than the nadir PSA achieved after SBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Kishan AU, Lamb JM, Wilhalme H, Casado M, Chong N, Zello L, Juarez JE, Jiang T, Neilsen BK, Low DA, Yang Y, Neylon J, Basehart V, Martin Ma T, Valle LF, Cao M, Steinberg ML. Magnetic Resonance Imaging Versus Computed Tomography Guidance for Stereotactic Body Radiotherapy in Prostate Cancer: 2-year Outcomes from the MIRAGE Randomized Clinical Trial. Eur Urol. 2025 Jun;87(6):622-625. doi: 10.1016/j.eururo.2024.10.026. Epub 2024 Nov 13. PMID 39537438
- [Derived] Kishan AU, Ma TM, Lamb JM, Casado M, Wilhalme H, Low DA, Sheng K, Sharma S, Nickols NG, Pham J, Yang Y, Gao Y, Neylon J, Basehart V, Cao M, Steinberg ML. Magnetic Resonance Imaging-Guided vs Computed Tomography-Guided Stereotactic Body Radiotherapy for Prostate Cancer: The MIRAGE Randomized Clinical Trial. JAMA Oncol. 2023 Mar 1;9(3):365-373. doi: 10.1001/jamaoncol.2022.6558. PMID 36633877
- [Derived] Ma TM, Lamb JM, Casado M, Wang X, Basehart TV, Yang Y, Low D, Sheng K, Agazaryan N, Nickols NG, Cao M, Steinberg ML, Kishan AU. Magnetic resonance imaging-guided stereotactic body radiotherapy for prostate cancer (mirage): a phase iii randomized trial. BMC Cancer. 2021 May 11;21(1):538. doi: 10.1186/s12885-021-08281-x. PMID 33975579